CLINICAL TRIAL: NCT07302503
Title: Pilot Study Evaluating brainQuant's Ability to Detect Alterations in White Matter in Diffusion MRI, Indicative of Post-traumatic Lesions
Acronym: BQ TC-foot
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9451
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chronic Traumatic Encephalopathy
Keywords: Chronic Traumatic Encephalopathy; Post-traumatic lesions; Neurodegenerative brain abnormalities; Professional soccer players
MeSH Terms: conditions — Chronic Traumatic Encephalopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic traumatic encephalopathy (CTE) is a neurodegenerative disease described in boxing, but also in contact sports such as American football.

Soccer, due to repeated headers, could also be associated, albeit to a lesser degree, with the development of this type of pathology.

Indeed, it has been shown that playing soccer can be accompanied by cognitive impairments, and neurodegenerative brain abnormalities have been described in neuropathology studies of former professional soccer players. Subradiological brain abnormalities have been found in multimodal MRI in various sports. Similarly, a decrease in cognitive performance has been described.

The discovery of this type of anomaly in a population of professional footballers nearing the end of their careers could lead to:

* The implementation of appropriate monitoring for professional footballers through early detection of lesions via MRI and cognitive disorders
* The implementation of preventative measures for professional footballers, but also for amateur footballers from a very young age.

ELIGIBILITY:
Inclusion Criteria:

* Male subject
* Aged 32 to 60 years inclusive
* Professional footballer nearing the end of their career or recently retired, or subject who has never regularly participated in sports that expose them to head trauma (particularly rugby, basketball, handball, American football, hockey, combat sports, etc.)

Exclusion Criteria:

- Subject who expressed their opposition to participating in the study

Ages: 32 Years to 60 Years | Sex: Male
Age Groups: Adult
Study Population: Male subject aged 32 to 60 years
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Changes found in MRI diffusion tensor imaging of professional football players | day 1 post-consultation

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Imagerie 2 - Réanimation - CHU de Strasbourg - France, Strasbourg, France